CLINICAL TRIAL: NCT01597388
Title: A Phase I, Open-label, Multicentre, Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of AZD2014 Administered Orally in Combination With Intramuscular (IM) Fulvestrant to Patients With Estrogen Receptor Positive (ER+) Advanced, Metastatic Breast Cancer
Brief Title: AZD2014 and Fulvestrant in Patients With ER+ Advanced Metastatic Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D2270C00005; BRE-196; 264477 (Other: Parexel International (IRL) Limited)
Record Dates: First submitted 2012-03-28; First posted 2012-05-14 (Estimated); Results first posted 2018-10-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Advanced Metastatic Breast Cancer
Keywords: Estrogen receptor positive; Advanced metastatic breast cancer; Estrogen receptor positive advanced metastatic breast cancer
MeSH Terms: interventions — vistusertib; Fulvestrant

ARMS (1):
- AZD2014 with Fulvestrant (Experimental): AZD2014 with Fulvestrant
  Interventions: Drug: AZD2014; Drug: Fulvestrant

INTERVENTIONS:
Drug: AZD2014 — Single dose followed by multiple dosing or twice daily dosing for 2 days folllowed by 5 days off each week, or twice daily dosing on the first and fourth day of the week
Drug: Fulvestrant — IM monthly after loading dose
  Other Names: faslodex

SUMMARY:
The purpose of this study is to assess safety and tolerability of AZD2014 when given in combination with Fulvestrant

DETAILED DESCRIPTION:
A Phase I, Open-label, Multicentre, Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of AZD2014 Administered Orally in Combination with Intramuscular (IM) Fulvestrant to Patients with Estrogen Receptor Positive (ER+) Advanced, Metastatic Breast Cancer.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated written informed consent prior to any study specific procedures, sampling analysis
* Aged at least 18
* At least one lesion (measurable and/or non-measurable) that can be accurately assessed at baseline by computerised tomography (CT) magnetic resonance imaging (MRI) or plain X-ray and is suitable for repeated assessment
* Histological or cytological confirmation of an ER+ advanced metastatic breast cancer tumour that is eligible for treatment with fulvestrant
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Patients must have evidence of non-child-bearing potential.

Exclusion Criteria:

* Prior chemotherapy, biological therapy, radiation therapy, androgens, thalidomide, immunotherapy, other anticancer agents, and any investigational agents within 14 days of starting study treatment (not including palliative radiotherapy at focal sites)
* Major surgery within 4 weeks prior to entry to the study (excluding placement of vascular access), or minor surgery within 2 weeks of entry into the study.
* Patients with severe cardiac condition of ischemia, impaired ventricular function and arrhythmias, evidence of severe or uncontrolled systemic or current unstable or uncompensated respiratory or cardiac conditions.
* Patients with diabetes type 1 or uncontrolled type II (HbA1c > 8% assessed locally)

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2012-05-08 (Actual); Primary Completion 2016-08-04 (Actual); Study Completion 2026-02-27 (Estimated)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Research Site, Sarasota, Florida
  - Research Site, Detroit, Michigan
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Greenville, South Carolina
  - Research Site, Nashville, Tennessee

REFERENCES:
- See also: AstraZeneca Cancer Study Locator Service http://www.emergingmed.com/networks/AstraZeneca astrazeneca@emergingmed.com 1-877-400-4656 — http://www.emergingmed.com/networks/AstraZeneca

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred ten (110) patients enrolled in the study; 100 patients were assigned to a treatment schedule and 10 patients were screen failures. One patient withdrew from the study prior to receiving study drug and was excluded from the safety analysis set.
  Patients were treated at 5 sites in the US from 21 May 2012 until 4 August 2016.
Groups:
- 35 mg BID Continuous: Participants took 35 mg of AZD2014 twice daily continuously in 28 day cycles. Participants also received intramuscular fulvestrant 500 mg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent cycle.
- 50 mg BID Continuous: Participants took 50 mg of AZD2014 twice daily continuously in 28 day cycles. Participants also received intramuscular fulvestrant 500 mg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent cycle.
- 75 mg QD Continuous: Participants took 75 mg of AZD2014 one time each day continuously in 28 day cycles. Participants also received intramuscular fulvestrant 500 mg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent cycles.
- 100 mg QD Continuous: Participants took 100 mg of AZD2014 one time each day continuously in 28 day cycles. Participants also received intramuscular fulvestrant 500 mg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent cycles.
- 125 mg BID Intermittent Days 1 and 2 (Fasted): Participants took 125 mg of AZD2014 twice daily on Days 1 and 2 of each week in 28 day cycles (4 weeks) in a fasted condition. Participants also received intramuscular fulvestrant 500 mg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent cycle.
- 125 mg BID Intermittent Days 1 and 2 (Fed): Participants took 125 mg of AZD2014 twice daily on Days 1 and 2 of each week in 28 day cycles (4 weeks) after eating. Participants also received intramuscular fulvestrant 500 mg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent cycle.
- 170 mg BID Intermittent Days 1 and 2 (Fasted): Participants took 170 mg of AZD2014 twice daily on Days 1 and 2 of each week in 28 day cycles (4 weeks) in a fasted condition. Participants also received intramuscular fulvestrant 500 mg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent cycle.
- 170 mg BID Intermittent Days 1 and 2 (Fed): Participants took 170 mg of AZD2014 twice daily on Days 1 and 2 of each week in 28 day cycles (4 weeks) after eating. Participants also received intramuscular fulvestrant 500 mg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent cycle.
- 125 mg BID Intermittent Days 1 and 4 (Fasted): Participants took 125 mg of AZD2014 twice daily on Days 1 and 4 of each week in 28 day cycles (4 weeks) in a fasted condition. Participants also received intramuscular fulvestrant 500 mg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent cycle.
Period: Overall Study
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous | 125 mg BID Intermittent Days 1 and 2 (Fasted) | 125 mg BID Intermittent Days 1 and 2 (Fed) | 170 mg BID Intermittent Days 1 and 2 (Fasted) | 170 mg BID Intermittent Days 1 and 2 (Fed) | 125 mg BID Intermittent Days 1 and 4 (Fasted)
Started | 6 | 13 | 14 | 10 | 37 | 4 | 8 | 5 | 2
Completed | 6 | 13 | 14 | 10 | 37 | 4 | 8 | 5 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 170 mg BID Intermittent Days 1 and 2 (Fasted): Participants took 170 mg of AZD2014 twice daily on Days 1 and 4 of each week in 28 day cycles (4 weeks) in a fasted condition. Participants also received intramuscular fulvestrant 500 mg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent cycle.
- Total: Total of all reporting groups
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous | 125 mg BID Intermittent Days 1 and 2 (Fasted) | 125 mg BID Intermittent Days 1 and 2 (Fed) | 170 mg BID Intermittent Days 1 and 2 (Fasted) | 170 mg BID Intermittent Days 1 and 2 (Fed) | 125 mg BID Intermittent Days 1 and 4 (Fasted) | Total
Number analyzed (Participants) | 6 | 13 | 14 | 10 | 37 | 4 | 8 | 5 | 2 | 99
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.5 (9.16) | 63.3 (12.53) | 61.1 (7.46) | 60.1 (10.46) | 60.1 (10.05) | 55.8 (6.29) | 54.4 (9.44) | 58.4 (9.26) | 55.0 (NA) — The standard deviation was not calculated because there were only 2 participants in this group. | 59.9 (9.88)
Age, Continuous [Median (Full Range); unit: Years] | 58.5 [48 to 72] | 64.0 [32 to 82] | 61.0 [50 to 76] | 62.0 [39 to 73] | 61.0 [40 to 77] | 55.0 [50 to 63] | 55.5 [34 to 64] | 59.0 [43 to 67] | 55.0 [43 to 67] | 61.0 [32 to 82]
Age, Customized [Count of Participants; unit: Participants]
  ≥18 and <50 years | 1 | 1 | 0 | 1 | 7 | 0 | 1 | 1 | 1 | 13
  ≥50 to <65 years | 3 | 6 | 8 | 5 | 18 | 4 | 7 | 3 | 0 | 54
  ≥65 years | 2 | 6 | 6 | 4 | 12 | 0 | 0 | 1 | 1 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 13 | 14 | 10 | 37 | 4 | 8 | 5 | 2 | 99
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 0 | 1 | 2 | 0 | 24 | 4 | 5 | 4 | 2 | 42
  Unknown or Not Reported | 6 | 12 | 12 | 9 | 13 | 0 | 3 | 1 | 0 | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 6 | 11 | 12 | 10 | 35 | 2 | 7 | 5 | 2 | 90
  Black or African American | 0 | 2 | 2 | 0 | 2 | 1 | 1 | 0 | 0 | 8
  Other | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 13 | 14 | 10 | 37 | 4 | 8 | 5 | 2 | 99
Weight [Mean (Standard Deviation); unit: kg] | 77.42 (15.953) | 73.29 (18.845) | 74.51 (19.236) | 74.53 (23.776) | 67.62 (15.511) | 79.88 (17.854) | 68.95 (14.115) | 77.98 (12.586) | 77.45 (NA) — The standard deviation was not calculated because there were only 2 participants in this arm. | 71.96 (17.134)
ECOG Performance Status (PS) [Count of Participants; unit: Participants] — ECOG PS = 0 Fully active; PS = 1 Restricted in physically strenuous activity; PS = 2 Ambulatory and capable of self-care; PS = Capable of only limited self care; PS = 4 Completely disabled
  Participants
    PS = 0 | 3 | 11 | 8 | 5 | 16 | 2 | 5 | 1 | 1 | 52
    PS = 1 | 3 | 2 | 6 | 5 | 21 | 2 | 3 | 4 | 1 | 47
    PS = 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    PS = 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    PS = 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour Grade [Count of Participants; unit: Participants] — G1 = Well differentiated; G2 = Moderately differentiated; G3 = Poorly differentiated; G4 = Undifferentiated; Gx = Not assessable
  Participants
    G1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 4
    G2 | 3 | 5 | 6 | 6 | 14 | 1 | 2 | 1 | 1 | 39
    G3 | 1 | 4 | 3 | 2 | 8 | 1 | 1 | 2 | 1 | 23
    G4 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
    Gx | 1 | 3 | 5 | 1 | 10 | 1 | 4 | 0 | 0 | 25
    Missing | 1 | 1 | 0 | 0 | 4 | 0 | 0 | 1 | 0 | 7
Histology Type [Count of Participants; unit: Participants]
  Cannot be determined | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Invasive carcinoma (NOS) | 0 | 1 | 1 | 1 | 4 | 1 | 0 | 0 | 0 | 8
  Invasive ductal | 4 | 6 | 7 | 5 | 17 | 1 | 5 | 4 | 1 | 50
  Invasive ductal/extensive intraductal component | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 4
  Invasive lobular | 2 | 3 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 9
  Other | 0 | 2 | 5 | 2 | 11 | 2 | 3 | 1 | 1 | 27
Malignant pleural effusion [Count of Participants; unit: Participants]
  Absent | 5 | 12 | 14 | 7 | 33 | 1 | 7 | 5 | 2 | 86
  Present | 1 | 1 | 0 | 3 | 4 | 3 | 1 | 0 | 0 | 13
Time from Diagnosis to Enrollment [Count of Participants; unit: Participants]
  ≤ 6 months | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  > 6 to ≤ 12 months | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  > 12 to ≤ 24 months | 0 | 1 | 0 | 1 | 4 | 0 | 0 | 0 | 0 | 6
  > 24 months | 6 | 12 | 13 | 9 | 33 | 4 | 8 | 5 | 2 | 92
Time from most recent progression to enrollment [Count of Participants; unit: Participants]
  ≤ 3 months | 5 | 11 | 12 | 8 | 28 | 3 | 8 | 5 | 2 | 82
  During screening, after informed consent | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  > 3 to ≤ 12 months | 0 | 1 | 2 | 2 | 5 | 1 | 0 | 0 | 0 | 11
  > 12 months | 0 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 4
Overall disease classification [Count of Participants; unit: Participants]
  Metastatic | 6 | 13 | 14 | 9 | 37 | 4 | 8 | 5 | 2 | 98
  Locally advanced | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Estrogen Receptor Positive (ER+) [Count of Participants; unit: Participants]
  Yes | 6 | 13 | 14 | 10 | 37 | 4 | 8 | 5 | 2 | 99
  No | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Progesterone Receptor Positive (PR+) [Count of Participants; unit: Participants]
  Yes | 3 | 7 | 7 | 7 | 30 | 4 | 4 | 1 | 2 | 65
  No | 3 | 6 | 7 | 3 | 7 | 0 | 4 | 4 | 0 | 34
Human Epidermal Growth Factor Receptor Positive (HER+) [Count of Participants; unit: Participants]
  Yes | 0 | 1 | 0 | 1 | 4 | 0 | 2 | 1 | 0 | 9
  No | 6 | 12 | 14 | 9 | 33 | 4 | 6 | 4 | 2 | 90

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events
Time Frame: Up to 12 Months
Population: The analysis population consisted of all participants who received at least one dose of AZD2014.
Measure: Number; unit: Participants
Groups:
- 75 mg QD Continuous: Participants took 75 mg of AZD2014 one time per day continuously in 28 day cycles. Participants also received intramuscular fulvestrant 500 mg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent cycle.
- 100 mg QD Continuous: Participants took 100 mg of AZD2014 one time per day in 28 day cycles (4 weeks). Participants also received intramuscular fulvestrant 500 mg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent cycle.
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous | 125 mg BID Intermittent Days 1 and 2 (Fasted) | 125 mg BID Intermittent Days 1 and 2 (Fed) | 170 mg BID Intermittent Days 1 and 2 (Fasted) | 170 mg BID Intermittent Days 1 and 2 (Fed) | 125 mg BID Intermittent Days 1 and 4 (Fasted)
Number analyzed (Participants) | 6 | 13 | 14 | 10 | 37 | 4 | 8 | 5 | 2
Participants
  Any Adverse Event (AE) | 6 | 13 | 14 | 10 | 37 | 4 | 8 | 5 | 2
  Any AE, Causally Related to AZD2014 | 5 | 12 | 14 | 9 | 35 | 4 | 8 | 5 | 2
  Any AE, Causally Related to Fulvestrant Only | 2 | 3 | 6 | 3 | 12 | 0 | 2 | 0 | 1
  Any AE of CTCAE Grade ≥ 3 (G3) | 3 | 8 | 10 | 6 | 24 | 3 | 6 | 3 | 1
  AEs of CTCAE G3, Causally Related to AZD2014 | 2 | 8 | 7 | 5 | 16 | 0 | 6 | 2 | 0
  Any AE of CTCAE G3, Related to Fulvestrant Only | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Adverse Event with Outcome of Death | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  AE with Outcome of Death, Related to AZD2014 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  AE Outcome of Death, Related to Fulvestrant Only | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Serious Adverse Event (SAE) | 0 | 1 | 3 | 1 | 7 | 0 | 3 | 1 | 0
  Any SAE, Causally Related to AZD2014 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 0
  Any SAE, Causally Related to Fulvestrant Only | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any AE Leading to Discontinuation of AZD2014 | 2 | 4 | 2 | 3 | 2 | 0 | 2 | 0 | 0
  Any SAE Leading to Discontinuation of AZD2014 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0

2. Primary Outcome: Adverse Events Leading to Dose Reduction of AZD2014
Time Frame: Up to 28 Days
Population: The analysis population consisted of all participants who received at least one dose of AZD2014.
Measure: Number; unit: Participants
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous | 125 mg BID Intermittent Days 1 and 2 (Fasted) | 125 mg BID Intermittent Days 1 and 2 (Fed) | 170 mg BID Intermittent Days 1 and 2 (Fasted) | 170 mg BID Intermittent Days 1 and 2 (Fed) | 125 mg BID Intermittent Days 1 and 4 (Fasted)
Number analyzed (Participants) | 6 | 13 | 14 | 10 | 37 | 4 | 8 | 5 | 2
Participants | 1 | 7 | 4 | 6 | 12 | 0 | 4 | 3 | 2

3. Primary Outcome: Clinically Important Changes in Haematology Parameters
Time Frame: Up to 12 Months
Population: The analysis population consisted of all participants who received at least one dose of AZD2014.
Measure: Number; unit: Participants
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous | 125 mg BID Intermittent Days 1 and 2 (Fasted) | 125 mg BID Intermittent Days 1 and 2 (Fed) | 170 mg BID Intermittent Days 1 and 2 (Fasted) | 170 mg BID Intermittent Days 1 and 2 (Fed) | 125 mg BID Intermittent Days 1 and 4 (Fasted)
Number analyzed (Participants) | 6 | 13 | 14 | 10 | 37 | 4 | 8 | 5 | 2
Participants
  Change in Hemoglobin ≥ 2 CTCAE Grades | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Change in Hemoglobin to CTCAE Grade 3 or 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Change in Leukocytes ≥ 2 CTCAE Grades | 0 | 4 | 2 | 1 | 9 | 2 | 2 | 3 | 0
  Change in Leukocytes to CTCAE Grade 3 or 4 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Change in Lymphocytes ≥ 2 CTCAE Grades | 2 | 6 | 8 | 5 | 10 | 0 | 1 | 2 | 1
  Change in Lymphocytes to CTCAE Grade 3 or 4 | 0 | 3 | 3 | 0 | 7 | 1 | 1 | 1 | 1
  Change in Neutrophils ≥ 2 CTCAE Grades | 1 | 4 | 1 | 3 | 12 | 1 | 1 | 1 | 0
  Change in Neutrophils to CTCAE Grade 3 or 4 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
  Change in Platelets ≥ 2 CTCAE Grades | 0 | 0 | 2 | 0 | 2 | 1 | 1 | 0 | 0
  Change in Platelets to CTCAE Grade 3 or 4 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
  Change in aPTT ≥ 2 CTCAE Grades | 0 | 1 | 0 | 0 | 3 | 0 | 1 | 1 | 0
  Change in aPTT to CTCAE Grade 3 or 4 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Change in INR ≥ 2 CTCAE Grades | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Change in INR to CTCAE Grade 3 or 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Clinically Important Changes in Clinical Chemistry Parameters
Time Frame: Up to 12 Months
Population: The analysis population consisted of all participants who received at least one dose of AZD2014.
Measure: Number; unit: Participants
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous | 125 mg BID Intermittent Days 1 and 2 (Fasted) | 125 mg BID Intermittent Days 1 and 2 (Fed) | 170 mg BID Intermittent Days 1 and 2 (Fasted) | 170 mg BID Intermittent Days 1 and 2 (Fed) | 125 mg BID Intermittent Days 1 and 4 (Fasted)
Number analyzed (Participants) | 6 | 13 | 14 | 10 | 37 | 4 | 8 | 5 | 2
Participants
  Change in ALT ≥ 2 CTCAE Grades | 0 | 1 | 3 | 3 | 0 | 1 | 0 | 0 | 0
  Change in ALT to CTCAE Grade 3 or 4 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0
  Change in AST ≥ 2 CTCAE Grades | 0 | 2 | 3 | 2 | 2 | 0 | 0 | 0 | 1
  Change in AST to CTCAE Grade 3 or 4 | 0 | 0 | 5 | 2 | 3 | 1 | 0 | 0 | 1
  Change in Alk Phosphatase ≥ 2 CTCAE Grades | 0 | 2 | 1 | 0 | 1 | 0 | 1 | 0 | 0
  Change in Alk Phosphatase to CTCAE Grade 3 or 4 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 0
  Change in Albumin ≥ 2 CTCAE Grades | 0 | 1 | 2 | 2 | 6 | 1 | 2 | 1 | 0
  Change in Albumin to CTCAE Grade 3 or 4 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Change in Bilirubin ≥ 2 CTCAE Grades | 1 | 0 | 1 | 0 | 3 | 0 | 2 | 1 | 0
  Change in Bilirubin to CTCAE Grade 3 or 4 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Change in Creatinine ≥ 2 CTCAE Grades | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0
  Change in Creatinine to CTCAE Grade 3 or 4 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Change in Phosphate ≥ 2 CTCAE Grades | 1 | 2 | 0 | 2 | 15 | 1 | 1 | 2 | 0
  Change in Phosphate to CTCAE Grade 3 or 4 | 0 | 0 | 0 | 0 | 7 | 0 | 0 | 1 | 0
  Change in Urate ≥ 2 CTCAE Grades | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Change in Urate to CTCAE Grade 3 or 4 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Change in Calcium ≥ 2 CTCAE Grades | 0 | 3 | 1 | 0 | 6 | 1 | 2 | 2 | 0
  Change in Calcium to CTCAE Grade 3 or 4 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0
  Change in Sodium ≥ 2 CTCAE Grades | 0 | 1 | 0 | 3 | 1 | 0 | 0 | 0 | 0
  Change in Sodium to CTCAE Grade 3 or 4 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
  Change in Potassium ≥ 2 CTCAE Grades | 1 | 1 | 2 | 5 | 5 | 1 | 0 | 0 | 0
  Change in Potassium to CTCAE Grade 3 or 4 | 0 | 0 | 1 | 5 | 5 | 1 | 0 | 0 | 0
  Change in Magnesium ≥ 2 CTCAE Grades | 0 | 1 | 0 | 2 | 1 | 0 | 2 | 0 | 0
  Change in Magnesium to CTCAE Grade 3 or 4 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0
  Change in Fasting Glucose ≥ 2 CTCAE Grades | 1 | 1 | 1 | 1 | 7 | 1 | 4 | 0 | 0
  Change in Fasting Glucose to CTCAE Grade 3 or 4 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0
  Change in NonFasting Glucose ≥ 2 CTCAE Grades | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2 | 0
  Change in Non Fasting Glucose to CTCAE Gr.3 or 4 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0

5. Primary Outcome: Left Ventricular Ejection Fraction
Time Frame: 24 hours
Population: The analysis population consisted of all participants who received at least one dose of AZD2014.
Measure: Mean (Standard Deviation); unit: % Left Ventricular Ejection Fraction
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous | 125 mg BID Intermittent Days 1 and 2 (Fasted) | 125 mg BID Intermittent Days 1 and 2 (Fed) | 170 mg BID Intermittent Days 1 and 2 (Fasted) | 170 mg BID Intermittent Days 1 and 2 (Fed) | 125 mg BID Intermittent Days 1 and 4 (Fasted)
Number analyzed (Participants) | 6 | 13 | 14 | 10 | 37 | 4 | 8 | 5 | 2
% Left Ventricular Ejection Fraction
  Screening | 59.2 (4.5) | 64.0 (5.4) | 60.9 (6.2) | 61.4 (9.8) | 62.6 (4.1) | 62.5 (2.9) | 66.9 (4.6) | 63.8 (5.2) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  End of Study | NA (NA) — Mean and SD were not calculated because data was available from < 3 participants. | 64.0 (2.0) | 62.3 (4.1) | 61.8 (8.3) | 62.5 (2.9) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  Change from Baseline to End of Study | NA (NA) — Mean and SD were not | 1.4 (5.9) | -1.5 (2.4) | 0.0 (7.6) | -1.3 (3.9) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.

6. Primary Outcome: QTcF Over 24 Hours
Time Frame: 24 hours
Population: The analysis population consisted of all participants who received at least one dose of AZD2014.
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous | 125 mg BID Intermittent Days 1 and 2 (Fasted) | 125 mg BID Intermittent Days 1 and 2 (Fed) | 170 mg BID Intermittent Days 1 and 2 (Fasted) | 170 mg BID Intermittent Days 1 and 2 (Fed) | 125 mg BID Intermittent Days 1 and 4 (Fasted)
Number analyzed (Participants) | 6 | 13 | 14 | 10 | 37 | 4 | 8 | 5 | 2
msec
  Baseline | 423.12 (11.070) | 421.92 (22.715) | 412.78 (14.222) | 415.95 (14.849) | 419.95 (20.502) | 427.13 (32.995) | 424.84 (6.932) | 435.26 (7.971) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  0.25 Hours Postdose | 429.66 (5.707) | 420.13 (18.333) | 413.04 (14.934) | 418.44 (16.145) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  0.5 Hours Postdose | 431.84 (7.504) | 419.18 (21.362) | 415.08 (14.762) | 418.91 (14.437) | 413.28 (19.715) | 418.90 (14.897) | 415.67 (16.874) | 420.06 (18.388) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  1 Hour Postdose | 431.00 (10.149) | 422.21 (21.863) | 416.08 (17.581) | 416.20 (14.530) | 416.22 (19.738) | 427.77 (10.186) | 419.61 (16.514) | 421.20 (21.336) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  1.5 Hours Postdose | 431.82 (8.569) | 425.15 (22.106) | 415.36 (16.394) | 415.33 (15.020) | 417.10 (19.672) | 434.33 (14.199) | 420.43 (15.627) | 427.48 (20.863) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  2 Hours Postdose | 433.02 (11.921) | 423.31 (22.678) | 415.84 (17.508) | 414.01 (17.988) | 414.99 (17.250) | 424.00 (22.528) | 418.60 (15.144) | 422.94 (18.036) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  4 Hours Postdose | 422.00 (10.583) | 419.97 (21.322) | 411.18 (15.886) | 410.88 (13.815) | 414.04 (17.351) | 424.43 (17.832) | 426.60 (16.724) | 422.40 (10.397) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  6 Hours Postdose | 421.50 (15.453) | 419.14 (21.269) | 411.85 (13.387) | 414.74 (16.413) | 412.80 (17.342) | 417.00 (20.421) | 422.94 (18.577) | 418.34 (13.781) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  8 Hours Postdose | 424.86 (12.688) | 420.16 (20.437) | 411.16 (15.587) | 413.56 (15.072) | 414.17 (18.533) | 419.90 (22.274) | 416.80 (15.144) | 425.54 (12.246) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  12 Hours Postdose | 427.74 (15.157) | 425.46 (21.533) | 409.67 (19.176) | 414.59 (15.760) | 414.09 (18.188) | 431.70 (16.896) | 420.66 (10.462) | 432.46 (16.503) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  24 Hours Postdose | 425.54 (10.519) | 421.45 (16.339) | 409.33 (16.313) | 415.29 (16.968) | 422.73 (17.900) | 426.77 (16.591) | NA (NA) — Data not collected | NA (NA) — Data not collected | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.

7. Primary Outcome: Post-Baseline Glucose Elevation
Time Frame: 28 Days
Population: The analysis population consisted of all participants who received at least one dose of AZD2014.
Measure: Number; unit: Participants
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous | 125 mg BID Intermittent Days 1 and 2 (Fasted) | 125 mg BID Intermittent Days 1 and 2 (Fed) | 170 mg BID Intermittent Days 1 and 2 (Fasted) | 170 mg BID Intermittent Days 1 and 2 (Fed) | 125 mg BID Intermittent Days 1 and 4 (Fasted)
Number analyzed (Participants) | 6 | 13 | 14 | 10 | 37 | 4 | 8 | 5 | 2
Participants
  Participants with ≥ 1 post-baseline elevation | 3 | 6 | 7 | 5 | 29 | 3 | 6 | 5 | 0
  Subjects with Max Post-Baseline CTCAE Grade ≥ 1 | 2 | 5 | 5 | 3 | 17 | 2 | 2 | 4 | 0
  Subjects with Max Post-Baseline CTCAE Grade ≥ 2 | 1 | 0 | 0 | 1 | 7 | 1 | 1 | 0 | 0
  Subjects with Max Post-Baseline CTCAE Grade ≥ 3 | 0 | 1 | 2 | 1 | 5 | 0 | 3 | 1 | 0
  Subjects with Max Post-Baseline CTCAE Grade ≥ 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Sitting Diastolic Blood Pressure
Time Frame: 28 Days
Population: The analysis population consisted of all participants who received at least one dose of AZD2014.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous | 125 mg BID Intermittent Days 1 and 2 (Fasted) | 125 mg BID Intermittent Days 1 and 2 (Fed) | 170 mg BID Intermittent Days 1 and 2 (Fasted) | 170 mg BID Intermittent Days 1 and 2 (Fed) | 125 mg BID Intermittent Days 1 and 4 (Fasted)
Number analyzed (Participants) | 6 | 13 | 14 | 10 | 37 | 4 | 8 | 5 | 2
mmHg
  Baseline | 72.8 (7.31) | 75.4 (10.43) | 77.4 (7.71) | 74.9 (8.36) | 74.4 (11.68) | 73.8 (8.62) | 75.5 (13.32) | 76.6 (8.59) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  Cycle 1, Day 1 | 74.8 (9.43) | 77.4 (9.82) | 75.4 (6.91) | 76.5 (8.03) | 74.4 (11.68) | 73.8 (8.62) | 75.5 (12.32) | 76.6 (8.59) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  Cycle 1, Day 8 | 74.5 (5.96) | 74.3 (8.58) | 75.3 (8.84) | 72.6 (12.68) | 72.4 (11.77) | 70.8 (5.38) | 78.3 (10.64) | 75.8 (7.63) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  Cycle 1, Day 15 | 74.7 (2.16) | 72.8 (8.64) | 75.4 (7.86) | 68.7 (7.12) | 73.1 (11.09) | 70.0 (7.87) | 74.2 (14.11) | 69.0 (9.59) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  Cycle 1, Day 22 | 72.5 (7.48) | 73.9 (9.37) | 76.2 (6.20) | 77.0 (5.40) | 70.9 (11.76) | 74.8 (10.24) | 75.0 (12.40) | 73.2 (13.10) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  Cycle 2, Day 1 | 72.0 (8.00) | 73.3 (10.49) | 72.7 (8.91) | 74.1 (7.36) | 71.4 (10.43) | 73.3 (4.57) | 72.5 (12.42) | 68.0 (5.29) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.

9. Primary Outcome: Sitting Systolic Blood Pressure
Time Frame: 28 Days
Population: The analysis population consisted of all participants who received at least one dose of AZD2014.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous | 125 mg BID Intermittent Days 1 and 2 (Fasted) | 125 mg BID Intermittent Days 1 and 2 (Fed) | 170 mg BID Intermittent Days 1 and 2 (Fasted) | 170 mg BID Intermittent Days 1 and 2 (Fed) | 125 mg BID Intermittent Days 1 and 4 (Fasted)
Number analyzed (Participants) | 6 | 13 | 14 | 10 | 37 | 4 | 8 | 5 | 2
mmHg
  Baseline | 114.2 (9.13) | 126.3 (14.65) | 127.4 (14.09) | 125.2 (20.82) | 124.4 (19.04) | 122.3 (14.31) | 120.8 (17.65) | 137.8 (19.18) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  Cycle 1, Day 1 | 113.5 (17.02) | 125.1 (15.68) | 122.6 (18.05) | 124.7 (14.51) | 124.4 (19.04) | 122.3 (14.31) | 120.8 (17.65) | 137.8 (19.18) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  Cycle 1, Day 8 | 124.0 (5.93) | 120.4 (9.12) | 123.7 (16.41) | 122.2 (20.67) | 122.2 (13.88) | 115.3 (13.30) | 127.9 (17.59) | 124.8 (21.56) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  Cycle 1, Day 15 | 119.7 (6.59) | 115.5 (17.50) | 121.6 (17.68) | 115.2 (9.17) | 122.8 (14.96) | 112.8 (13.10) | 128.3 (15.87) | 126.6 (10.97) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  Cycle 1, Day 22 | 116.7 (12.09) | 124.7 (16.92) | 123.5 (21.17) | 125.4 (16.67) | 116.6 (16.62) | 115.5 (15.50) | 119.9 (19.18) | 109.2 (8.32) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  Cycle 2, Day 1 | 111.7 (17.83) | 119.7 (17.59) | 123.6 (24.89) | 116.6 (10.31) | 119.3 (17.81) | 112.5 (9.00) | 113.2 (18.54) | 117.0 (9.06) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.

10. Primary Outcome: Respiratory Rate
Time Frame: 28 Days
Population: The analysis population consisted of all participants who received at least one dose of AZD2014.
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous | 125 mg BID Intermittent Days 1 and 2 (Fasted) | 125 mg BID Intermittent Days 1 and 2 (Fed) | 170 mg BID Intermittent Days 1 and 2 (Fasted) | 170 mg BID Intermittent Days 1 and 2 (Fed) | 125 mg BID Intermittent Days 1 and 4 (Fasted)
Number analyzed (Participants) | 6 | 13 | 14 | 10 | 37 | 4 | 8 | 5 | 2
breaths/min
  Baseline | 18.3 (2.66) | 17.5 (1.85) | 18.3 (1.33) | 17.8 (2.39) | 17.5 (0.96) | 17.5 (0.58) | 18.1 (0.83) | 17.6 (0.89) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  Cycle 1, Day 1 | 16.0 (1.63) | 16.6 (1.43) | 17.7 (1.33) | 17.3 (1.34) | 17.5 (0.96) | 17.5 (0.58) | 18.1 (0.83) | 17.6 (0.89) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  Cycle 1, Day 8 | 17.3 (1.63) | 16.4 (1.89) | 17.6 (1.34) | 17.5 (0.85) | 17.2 (1.47) | 16.8 (0.96) | 17.3 (1.89) | 18.0 (0.00) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  Cycle 1, Day 15 | 17.2 (0.98) | 17.1 (1.38) | 18.5 (1.20) | 17.9 (1.66) | 17.6 (1.03) | 17.0 (0.82) | 17.7 (0.82) | 17.4 (0.89) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  Cycle 1, Day 22 | 17.3 (2.07) | 17.8 (1.03) | 18.0 (1.15) | 17.1 (1.07) | 17.6 (1.54) | 17.8 (1.26) | 17.6 (0.79) | 18.0 (0.00) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  Cycle 2, Day 1 | 17.3 (1.63) | 17.6 (1.16) | 17.8 (0.99) | 18.3 (1.28) | 17.3 (2.11) | 17.8 (1.26) | 17.3 (1.03) | 17.5 (1.00) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.

11. Primary Outcome: Heart Rate
Time Frame: 28 Days
Population: The analysis population consisted of all participants who received at least one dose of AZD2014.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous | 125 mg BID Intermittent Days 1 and 2 (Fasted) | 125 mg BID Intermittent Days 1 and 2 (Fed) | 170 mg BID Intermittent Days 1 and 2 (Fasted) | 170 mg BID Intermittent Days 1 and 2 (Fed) | 125 mg BID Intermittent Days 1 and 4 (Fasted)
Number analyzed (Participants) | 6 | 13 | 14 | 10 | 37 | 4 | 8 | 5 | 2
beats/min
  Baseline | 87.5 (11.36) | 84.5 (13.31) | 82.7 (14.14) | 81.0 (13.11) | 83.5 (15.32) | 73.5 (10.75) | 86.1 (21.40) | 79.6 (5.32) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  Cycle 1, Day 1 | 87.3 (4.92) | 77.7 (14.28) | 87.3 (19.53) | 86.8 (12.90) | 83.5 (15.32) | 73.5 (10.75) | 86.1 (21.40) | 79.6 (5.32) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  Cycle 1, Day 8 | 80.8 (11.39) | 81.2 (15.93) | 85.4 (19.97) | 92.6 (12.47) | 84.4 (15.61) | 71.5 (6.61) | 79.4 (15.78) | 75.5 (12.01) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  Cycle 1, Day 15 | 80.2 (9.97) | 89.3 (16.83) | 86.7 (18.48) | 82.8 (8.60) | 81.3 (14.79) | 83.3 (15.33) | 82.5 (17.65) | 77.4 (7.92) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  Cycle 1, Day 22 | 82.4 (13.58) | 87.8 (16.95) | 85.3 (20.23) | 86.1 (11.18) | 84.6 (17.27) | 77.8 (7.80) | 87.4 (25.97) | 88.8 (11.43) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.
  Cycle 2, Day 1 | 83.5 (11.81) | 89.7 (11.63) | 84.0 (16.39) | 87.9 (12.45) | 85.7 (15.53) | 78.0 (15.75) | 83.0 (13.94) | 85.0 (12.68) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm.

12. Primary Outcome: Body Temperature
Time Frame: 28 Days
Population: The analysis population consisted of all participants who received at least one dose of AZD2014.
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous | 125 mg BID Intermittent Days 1 and 2 (Fasted) | 125 mg BID Intermittent Days 1 and 2 (Fed) | 170 mg BID Intermittent Days 1 and 2 (Fasted) | 170 mg BID Intermittent Days 1 and 2 (Fed) | 125 mg BID Intermittent Days 1 and 4 (Fasted)
Number analyzed (Participants) | 6 | 13 | 14 | 10 | 37 | 4 | 8 | 5 | 2
°C
  Baseline | 36.35 (0.327) | 36.44 (0.399) | 36.46 (0.303) | 36.48 (0.297) | 36.57 (0.320) | 36.60 (0.183) | 36.39 (0.482) | 36.40 (0.394) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm
  Cycle 1, Day 1 | 36.33 (0.189) | 36.57 (0.465) | 36.34 (0.318) | 36.46 (0.306) | 36.57 (0.320) | 36.60 (0.183) | 36.39 (0.482) | 36.40 (0.394) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm
  Cycle 1, Day 8 | 36.33 (0.308) | 36.42 (0.217) | 36.59 (0.493) | 36.35 (0.372) | 36.51 (0.370) | 36.25 (0.129) | 36.36 (0.276) | 36.88 (0.359) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm
  Cycle 1, Day 15 | 36.48 (0.313) | 36.74 (0.323) | 36.45 (0.333) | 36.35 (0.299) | 36.50 (0.400) | 36.30 (0.216) | 36.77 (0.489) | 36.42 (0.130) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm
  Cycle 1, Day 22 | 36.13 (0.403) | 36.38 (0.360) | 36.38 (0.414) | 36.26 (0.450) | 36.54 (0.550) | 36.65 (0.465) | 36.66 (0.341) | 36.88 (0.319) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm
  Cycle 2, Day 1 | 36.25 (0.315) | 36.55 (0.238) | 36.57 (0.312) | 36.54 (0.444) | 36.56 (0.292) | 36.90 (0.294) | 36.50 (0.456) | 36.54 (0.152) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm

13. Primary Outcome: Oxygen Saturation
Time Frame: 28 Days
Population: The analysis population consisted of all participants who received at least one dose of AZD2014.
Measure: Mean (Standard Deviation); unit: % Arterial Oxygen Saturation
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous | 125 mg BID Intermittent Days 1 and 2 (Fasted) | 125 mg BID Intermittent Days 1 and 2 (Fed) | 170 mg BID Intermittent Days 1 and 2 (Fasted) | 170 mg BID Intermittent Days 1 and 2 (Fed) | 125 mg BID Intermittent Days 1 and 4 (Fasted)
Number analyzed (Participants) | 6 | 13 | 14 | 10 | 37 | 4 | 8 | 5 | 2
% Arterial Oxygen Saturation
  Baseline | 97.0 (0.89) | 97.2 (1.59) | 96.8 (1.85) | 96.7 (2.41) | 97.8 (1.49) | 97.0 (1.83) | 97.0 (0.93) | 97.6 (1.14) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm
  Cycle 1, Day 1 | 97.5 (1.00) | 97.7 (1.90) | 97.4 (1.16) | 96.9 (1.90) | 97.8 (1.49) | 97.0 (1.83) | 97.0 (0.93) | 97.6 (1.14) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm
  Cycle 1, Day 8 | 98.3 (1.21) | 97.5 (1.98) | 97.1 (1.66) | 97.1 (1.37) | 97.8 (1.70) | 97.0 (2.16) | 97.7 (1.50) | 98.3 (2.06) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm
  Cycle 1, Day 15 | 97.7 (0.82) | 96.5 (1.94) | 97.3 (1.50) | 97.1 (1.17) | 98.0 (1.34) | 97.0 (1.41) | 97.0 (1.26) | 96.8 (1.48) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm
  Cycle 1, Day 22 | 96.8 (1.72) | 97.3 (1.82) | 96.8 (1.77) | 97.6 (1.51) | 98.1 (1.63) | 97.5 (3.11) | 97.9 (1.57) | 98.0 (1.63) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm
  Cycle 2, Day 1 | 97.5 (0.55) | 97.3 (2.09) | 96.9 (1.26) | 97.3 (1.04) | 98.2 (1.39) | 96.5 (2.52) | 96.2 (3.31) | 97.0 (2.16) | NA (NA) — Mean and standard deviation were not calculated because there were < 3 participants in this arm

14. Primary Outcome: AZD2014 Peak Plasma Concentration at Steady State (Cmax,ss) on Cycle 0 Days -5 to -1, Continuous Dosing, no Fulvestrant
Time Frame: 5 Days
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 35 mg BID Continuous: Participants took 35 mg of AZD2014 twice daily continuously in Cycle 0 on Days -5 to -1.
- 50 mg BID Continuous: Participants took 50 mg of AZD2014 twice daily continuously in Cycle 0 on Days -5 to -1.
- 75 mg QD Continuous: Participants took 75 mg of AZD2014 one time each day continuously in Cycle 0 on Days -5 to -1.
- 100 mg QD Continuous: Participants took 100 mg of AZD2014 one time each day continuously in Cycle 0 on Days -5 to -1.
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous
Number analyzed (Participants) | 5 | 13 | 14 | 10
ng/mL | 971.2 (413.6) | 1023 (339.4) | 1895 (965.6) | 2166 (964.3)

15. Primary Outcome: AZD2014 Area Under the Plasma Concentration Time Curve (AUC 0-12) Cycle 0 Days -5 to -1, Continuous Dosing, no Fulvestrant
Time Frame: 5 Days
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous
Number analyzed (Participants) | 5 | 13 | 14 | 10
h*ng/mL | 3478 (1398) | 5080 (1985) | 9723 (6408) | 12590 (4900)

16. Primary Outcome: AZD2014 Area Under the Plasma Concentration Time Curve (AUC 0-24) Cycle 0 Days -5 to -1, Continuous Dosing, no Fulvestrant
Time Frame: 5 Days
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous
Number analyzed (Participants) | 5 | 13 | 14 | 10
h*ng/mL | 3697 (1426) | 6006 (2838) | 11650 (8685) | 15790 (7286)

17. Primary Outcome: AZD2014 Area Under the Plasma Concentration Time Curve (AUC 0-t) Cycle 0 Days -5 to -1, Continuous Dosing, no Fulvestrant
Time Frame: 5 Days
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous
Number analyzed (Participants) | 5 | 13 | 14 | 10
h*ng/mL | 3458 (1433) | 5832 (2926) | 11500 (8761) | 15660 (7345)

18. Primary Outcome: AZD2014 Area Under the Plasma Concentration Time Curve (AUC 0-∞) Cycle 0 Days -5 to -1, Continuous Dosing, no Fulvestrant
Time Frame: 5 Days
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous
Number analyzed (Participants) | 5 | 13 | 14 | 10
h*ng/mL | 3731 (1412) | 6392 (3350) | 12360 (9950) | 17360 (9479)

19. Primary Outcome: AZD2014 Peak Plasma Concentration at Steady State (Cmax,ss) on Cycle 1 Day 15, BID Intermittent Dosing, With Fulvestrant
Time Frame: 15 Days
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 125 mg BID Intermittent Days 1 and 2 (Fasted) | 125 mg BID Intermittent Days 1 and 2 (Fed) | 170 mg BID Intermittent Days 1 and 2 (Fasted) | 170 mg BID Intermittent Days 1 and 2 (Fed)
Number analyzed (Participants) | 33 | 3 | 6 | 5
ng/mL | 3165 (1052) | 1933 (793.9) | 4238 (1440) | 2454 (838.4)

20. Primary Outcome: Time to AZD2014 Peak Plasma Concentration at Steady State (Tmax,ss) on Cycle 1 Day 15, BID Intermittent Dosing, With Fulvestrant
Time Frame: 15 Days
Measure: Median (Full Range); unit: hours
Arm/Group | 125 mg BID Intermittent Days 1 and 2 (Fasted) | 125 mg BID Intermittent Days 1 and 2 (Fed) | 170 mg BID Intermittent Days 1 and 2 (Fasted) | 170 mg BID Intermittent Days 1 and 2 (Fed)
Number analyzed (Participants) | 33 | 3 | 6 | 5
hours | 1.1 (1052) [0.5 to 4] | 2.0 (793.9) [1.07 to 6.15] | 1.5 (1440) [0.5 to 8] | 3.0 (838.4) [1 to 4]

21. Primary Outcome: AZD2014 Area Under the Plasma Concentration Time Curve (AUC 0-12) Cycle 1 Day 15 Intermittent Dosing, With Fulvestrant
Time Frame: 15 Days
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | 125 mg BID Intermittent Days 1 and 2 (Fasted) | 125 mg BID Intermittent Days 1 and 2 (Fed) | 170 mg BID Intermittent Days 1 and 2 (Fasted) | 170 mg BID Intermittent Days 1 and 2 (Fed)
Number analyzed (Participants) | 5 | 13 | 14 | 10
h*ng/mL | 19810 (6562) | 13760 (5737) | 26570 (8600) | 16150 (5591)

22. Primary Outcome: AZD2014 Peak Plasma Concentration at Steady State (Cmax,ss) on Cycle 1 Day 22, Continuous Dosing, With Fulvestrant
Time Frame: 22 Days
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- 75 mg QD Continuous; 100 mg QD Continuously: Participants took 100 mg of AZD2014 one time per day continuously in 28 day cycles (4 weeks). Participants also received intramuscular fulvestrant 500 mg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent cycle.
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuously
Number analyzed (Participants) | 6 | 10 | 11 | 6
ng/mL | 1374 (447.9) | 1785 (866) | 2409 (1305) | 2327 (1257)

23. Primary Outcome: Time to AZD2014 Peak Plasma Concentration at Steady State (Tmax,ss) on Cycle 1 Day 22, Continuous Dosing, With Fulvestrant
Time Frame: 22 Days
Measure: Median (Full Range); unit: hours
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuously
Number analyzed (Participants) | 6 | 10 | 11 | 6
hours | 1.3 (447.9) [0.5 to 4] | 1.0 (866) [0.5 to 2] | 1.5 (1305) [0.5 to 6.12] | 1.5 (1257) [0.5 to 6]

24. Primary Outcome: AZD2014 Area Under the Plasma Concentration Time Curve (AUC 0-12) Cycle 1 Day 22 Continuous Dosing, With Fulvestrant
Time Frame: 15 Days
Measure: Mean (Standard Deviation); unit: h*ng/mL
Groups:
- 35 mg BID Continuous: Participants took 35 mg of AZD2014 twice daily continuously in 28 day cycles (4 weeks). Participants also received intramuscular fulvestrant 500 mg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent cycle.
- 50 mg BID Continuous: Participants took 50 mg of AZD2014 twice daily continuously in 28 day cycles (4 weeks). Participants also received intramuscular fulvestrant 500 mg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent cycle.
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous
Number analyzed (Participants) | 6 | 10 | 11 | 6
h*ng/mL | 8611 (3864) | 11810 (7107) | 13510 (8937) | 15580 (6024)

25. Secondary Outcome: AZD2014 Peak Plasma Concentration (Cmax) Following Single Dose, Fasted, no Fulvestrant.
Time Frame: 1 Day
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- 35 mg: Participants received a single dose of 35 mg of AZD2014 in fasted condition.
- 50 mg: Participants received a single dose of 50 mg of AZD2014 in fasted condition.
- 75 mg: Participants received a single dose of 75 mg of AZD2014 in fasted condition.
- 100 mg: Participants received a single dose of 100 mg of AZD2014 in fasted condition.
Arm/Group | 35 mg | 50 mg | 75 mg | 100 mg
Number analyzed (Participants) | 5 | 13 | 14 | 10
ng/mL | 889.4 (52.72) | 968.5 (36.45) | 1678 (55.72) | 1942 (56.46)

26. Secondary Outcome: Time to AZD2014 Peak Plasma Concentration (Tmax) Following Single Dose, Fasted, no Fulvestrant.
Time Frame: 1 Day
Measure: Median (Full Range); unit: hour
Arm/Group | 35 mg | 50 mg | 75 mg | 100 mg
Number analyzed (Participants) | 5 | 13 | 14 | 10
hour | 1.00 (52.72) [0.50 to 1.50] | 1.00 (36.45) [0.45 to 4.00] | 1.10 (55.72) [0.50 to 4.00] | 1.80 (56.46) [0.50 to 4.02]

27. Secondary Outcome: Area Under the Plasma Concentration-time Curve for AZD2014 From 0 to 12 Hours (AUC 0-12) Following Single Dose, Fasted, no Fulvestrant.
Time Frame: 1 Day
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 35 mg | 50 mg | 75 mg | 100 mg
Number analyzed (Participants) | 5 | 13 | 14 | 10
h*ng/mL | 3233 (46.26) [0.50 to 1.50] | 4666 (48.2) [0.45 to 4.00] | 8185 (65.21) [0.50 to 4.00] | 11470 (53.45) [0.50 to 4.02]

28. Secondary Outcome: Area Under the Plasma Concentration-time Curve for AZD2014 From 0 to Infinity (AUC 0-∞) Following Single Dose, Fasted, no Fulvestrant.
Time Frame: 1 Day
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | 35 mg | 50 mg | 75 mg | 100 mg
Number analyzed (Participants) | 5 | 13 | 14 | 10
h*ng/mL | 3494 (43.96) [0.50 to 1.50] | 5543 (63.41) [0.45 to 4.00] | 9843 (75.43) [0.50 to 4.00] | 15110 (63.32) [0.50 to 4.02]

29. Secondary Outcome: Objective Response Rate
Description: Objective Response Rate (ORR) is defined as the number (%) of patients with a confirmed overall response of either complete response (CR) or partial response (PR).
Time Frame: Up to 12 months
Population: The population consisted of all patients receiving at least one dose of AZD 2014 and fulvestrant with measurable disease at baseline per RECIST v1.1.
Measure: Number; unit: Participants
Groups:
- 100 mg QD Continuous: Participants took 100 mg of AZD2014 one time per day continuously in 28 day cycles. Participants also received intramuscular fulvestrant 500 mg on Days 1 and 15 of Cycle 1 and on Day 1 of each subsequent cycle.
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous | 125 mg BID Intermittent Days 1 and 2 (Fasted) | 125 mg BID Intermittent Days 1 and 2 (Fed) | 170 mg BID Intermittent Days 1 and 2 (Fasted) | 170 mg BID Intermittent Days 1 and 2 (Fed) | 125 mg BID Intermittent Days 1 and 4 (Fasted)
Number analyzed (Participants) | 2 | 11 | 13 | 4 | 27 | 3 | 5 | 3 | 1
Participants | 0 | 2 | 2 | 1 | 2 | 1 | 1 | 0 | 1

30. Secondary Outcome: Best Objective Response (BOR)
Description: Best objective response was the best response a patient had following start of treatment but prior to starting any subsequent cancer therapy and prior to RECIST v1.1 progression or the last evaluable assessment in the absence of RECIST v1.1 progression.
Time Frame: Up to 12 months
Population: as for outcome 29
Measure: Number; unit: Participants
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous | 125 mg BID Intermittent Days 1 and 2 (Fasted) | 125 mg BID Intermittent Days 1 and 2 (Fed) | 170 mg BID Intermittent Days 1 and 2 (Fasted) | 170 mg BID Intermittent Days 1 and 2 (Fed) | 125 mg BID Intermittent Days 1 and 4 (Fasted)
Number analyzed (Participants) | 2 | 11 | 13 | 4 | 27 | 3 | 5 | 3 | 1
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 2 | 2 | 1 | 2 | 1 | 1 | 0 | 1
  Stable Disease ≥ 8 weeks | 1 | 4 | 7 | 1 | 17 | 2 | 3 | 1 | 0
  Progression | 1 | 2 | 3 | 0 | 7 | 0 | 0 | 1 | 0
  Not Evaluable | 0 | 3 | 1 | 2 | 1 | 0 | 1 | 1 | 0

31. Secondary Outcome: Duration of Response (DoR)
Description: Duration of response is defined as the time from the date of first documented response until the date of documented progression or death in the absence of disease progression.
Time Frame: Up to 12 months
Population: The number of participants analyzed for Duration of Response is zero in cohorts which had no responders [35 mg BID Continuous and 170 mg BID Intermittent Days 1 and 2 (fed)]
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous | 125 mg BID Intermittent Days 1 and 2 (Fasted) | 125 mg BID Intermittent Days 1 and 2 (Fed) | 170 mg BID Intermittent Days 1 and 2 (Fasted) | 170 mg BID Intermittent Days 1 and 2 (Fed) | 125 mg BID Intermittent Days 1 and 4 (Fasted)
Number analyzed (Participants) | 0 | 2 | 2 | 1 | 2 | 1 | 1 | 0 | 1
Months |  | 5.1 [3.9 to 6.3] | 9.7 [3.3 to 16.0] | NA [NA to NA] — Median and interquartile range can not be calculated because there was only one participant in the cohort. | NA [3.6 to NA] — Median and upper limit of the interquartile range can not be calculated for Duration of Response because response was ongoing for one participant at the time of data cut-off. | NA [NA to NA] — Median and interquartile range can not be calculated because there was only one participant in the cohort. | NA [NA to NA] — Median and interquartile range can not be calculated because there was only one participant in the cohort. |  | 10.4 [NA to NA] — Median and interquartile range can not be calculated because there was only one participant in the cohort.

32. Secondary Outcome: Clinical Benefit Rate (CBR) at 24 Weeks
Description: The Clinical Benefit Rate (CBR) at 24 weeks is defined as the percentage of patients who had a confirmed BOR of CR or PR in the first 24 weeks or who demonstrated SD for a minimum interval of 24 weeks (minus 1 week to allow for an early assessment within the assessment window, i.e., 161 days) following the start of treatment.
Time Frame: Up to 12 months
Population: The "tumour assessment" analysis set consisted of all participants who received at least one dose of AZD2014 and fulvestrant and had a baseline tumour assessment.
Measure: Number; unit: Participants
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous | 125 mg BID Intermittent Days 1 and 2 (Fasted) | 125 mg BID Intermittent Days 1 and 2 (Fed) | 170 mg BID Intermittent Days 1 and 2 (Fasted) | 170 mg BID Intermittent Days 1 and 2 (Fed) | 125 mg BID Intermittent Days 1 and 4 (Fasted)
Number analyzed (Participants) | 6 | 13 | 14 | 10 | 37 | 8 | 5 | 5 | 2
Participants
  Yes | 2 | 6 [3.6 to 6.3] | 4 [3.3 to 16.0] | 7 [39.1 to 39.1] | 11 [3.6 to NA] | 2 [6.4 to 6.4] | 3 [12.0 to 12.0] | 2 | 2 [10.4 to 10.4]
  No | 4 | 7 | 10 | 3 | 26 | 2 | 5 | 3 | 0

33. Secondary Outcome: Percentage Change From Baseline at 16 Weeks in Target Lesion (TL) Size.
Description: Baseline was defined as last evaluable assessment prior to starting treatment. Tumour size was the sum of the longest diameters of the target lesions. TLs are measurable tumour lesions.
Time Frame: Up to 12 months
Population: The "evaluable for response" analysis set consisted of all participants who received at least one dose of AZD2014 and fulvestrant and had measurable disease at baseline per RECIST v1.1.
Measure: Mean (Standard Deviation); unit: Percentage Change
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous | 125 mg BID Intermittent Days 1 and 2 (Fasted) | 125 mg BID Intermittent Days 1 and 2 (Fed) | 170 mg BID Intermittent Days 1 and 2 (Fasted) | 170 mg BID Intermittent Days 1 and 2 (Fed) | 125 mg BID Intermittent Days 1 and 4 (Fasted)
Number analyzed (Participants) | 2 | 10 | 12 | 2 | 26 | 3 | 5 | 2 | 1
Percentage Change | NA (NA) — Mean change in tumour size and standard deviation are not reported when data are available for less than 3 patients. | -9.37 (39.544) | -5.83 (52.781) | NA (NA) — Mean change in tumour size and standard deviation are not reported when data are available for less than 3 patients. | -0.46 (28.208) | -3.57 (28.476) | -10.96 (19.012) | NA (NA) — Mean change in tumour size and standard deviation are not reported when data are available for less than 3 patients. | NA (NA) — Mean change in tumour size and standard deviation are not reported when data are available for less than 3 patients.

34. Secondary Outcome: Progression Free Survival
Time Frame: Up to 12 months
Population: as for outcome 32
Measure: Median (80% Confidence Interval); unit: Weeks
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous | 125 mg BID Intermittent Days 1 and 2 (Fasted) | 125 mg BID Intermittent Days 1 and 2 (Fed) | 170 mg BID Intermittent Days 1 and 2 (Fasted) | 170 mg BID Intermittent Days 1 and 2 (Fed) | 125 mg BID Intermittent Days 1 and 4 (Fasted)
Number analyzed (Participants) | 6 | 13 | 14 | 10 | 37 | 4 | 8 | 5 | 2
Weeks | 49.4 (NA) [8.14 to 82.86] | 35.6 (39.544) [25.57 to 44.43] | 17.3 (52.781) [16.00 to 21.00] | 78.3 (NA) [57.00 to 178.14] | 22.6 (28.208) [16.14 to 25.14] | 33.9 (28.476) [17.14 to NA] — The upper bound of the 80% C.I. was not a finite number | 60.1 (19.012) [16.00 to NA] — The upper bound of the 80% C.I. was not a finite number | 83.4 (NA) [7.14 to 83.43] | NA (NA) [61.86 to NA] — The median could not be determined because only 1 progression event occurred in this arm. The upper bound of the 80% C.I. was not a finite number

35. Secondary Outcome: Progression Free Survival at 26 Weeks
Time Frame: Up to 12 months
Population: as for outcome 32
Measure: Number (80% Confidence Interval); unit: Percentage
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous | 125 mg BID Intermittent Days 1 and 2 (Fasted) | 125 mg BID Intermittent Days 1 and 2 (Fed) | 170 mg BID Intermittent Days 1 and 2 (Fasted) | 170 mg BID Intermittent Days 1 and 2 (Fed) | 125 mg BID Intermittent Days 1 and 4 (Fasted)
Number analyzed (Participants) | 6 | 13 | 14 | 10 | 37 | 4 | 8 | 5 | 2
Percentage | 33 (NA) [9.3 to 66.7] | 38 (39.544) [20.1 to 59.8] | 21 (52.781) [8.1 to 41.7] | 60 (NA) [35.4 to 81.2] | 35 (28.208) [24.6 to 47.0] | 50 (28.476) [14.3 to 85.7] | 38 (19.012) [14.7 to 65.5] | 40 (NA) [11.2 to 75.3] | 100 (NA) [31.6 to 100.0]

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | 35 mg BID Continuous | 50 mg BID Continuous | 75 mg QD Continuous | 100 mg QD Continuous | 125 mg BID Intermittent Days 1 and 2 (Fasted) | 125 mg BID Intermittent Days 1 and 2 (Fed) | 170 mg BID Intermittent Days 1 and 2 (Fasted) | 170 mg BID Intermittent Days 1 and 2 (Fed) | 125 mg BID Intermittent Days 1 and 4 (Fasted)
Serious Adverse Events (participants affected / at risk) | 0/6 | 1/13 | 3/14 | 1/10 | 7/37 | 0/4 | 3/8 | 1/5 | 0/2
Other Adverse Events (participants affected / at risk) | 6/6 | 13/13 | 14/14 | 10/10 | 37/37 | 4/4 | 8/8 | 5/5 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 35 mg BID Continuous (N=6) | 50 mg BID Continuous (N=13) | 75 mg QD Continuous (N=14) | 100 mg QD Continuous (N=10) | 125 mg BID Intermittent Days 1 and 2 (Fasted) (N=37) | 125 mg BID Intermittent Days 1 and 2 (Fed) (N=4) | 170 mg BID Intermittent Days 1 and 2 (Fasted) (N=8) | 170 mg BID Intermittent Days 1 and 2 (Fed) (N=5) | 125 mg BID Intermittent Days 1 and 4 (Fasted) (N=2)
Evans Syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascities (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 35 mg BID Continuous (N=6) | 50 mg BID Continuous (N=13) | 75 mg QD Continuous (N=14) | 100 mg QD Continuous (N=10) | 125 mg BID Intermittent Days 1 and 2 (Fasted) (N=37) | 125 mg BID Intermittent Days 1 and 2 (Fed) (N=4) | 170 mg BID Intermittent Days 1 and 2 (Fasted) (N=8) | 170 mg BID Intermittent Days 1 and 2 (Fed) (N=5) | 125 mg BID Intermittent Days 1 and 4 (Fasted) (N=2)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 3 (4) | 1 (1) | 3 (4) | 0 (0) | 2 (2) | 0 (0) | 1 (2)
Anaemia of Malignant Disease (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (8) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain, Upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (3) | 1 (1) | 11 (11) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 8 (8) | 7 (10) | 5 (8) | 19 (26) | 0 (0) | 7 (12) | 1 (1) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (3) | 5 (5) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 6 (7) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 7 (9) | 7 (8) | 9 (15) | 28 (39) | 3 (3) | 8 (15) | 3 (4) | 2 (2)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 8 (11) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 3 (4) | 9 (12) | 6 (6) | 7 (10) | 13 (16) | 1 (1) | 4 (6) | 2 (6) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (5) | 4 (5) | 3 (4) | 19 (29) | 3 (5) | 8 (18) | 3 (4) | 1 (1)
Asthenia (General disorders) | 0 (0) | 2 (2) | 3 (3) | 2 (3) | 10 (10) | 1 (1) | 4 (4) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3/3 (3) | 7 (13) | 9 (10) | 7 (10) | 23 (24) | 3 (4) | 5 (6) | 4 (5) | 2 (2)
Oedema Peripheral (General disorders) | 1 (1) | 3 (5) | 6 (8) | 0 (0) | 7 (7) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (4) | 3 (3) | 4 (4) | 6 (8) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 2 (3) | 8 (10) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (4) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 8 (9) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Blood Creatinine Increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breath Sounds Abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (5) | 0 (0) | 0 (0)
Transaminases Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Weight Decreased (Investigations) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 10 (10) | 2 (2) | 2 (2) | 3 (3) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 5 (5) | 3 (3) | 4 (4) | 15 (16) | 1 (1) | 3 (4) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 4 (5) | 2 (2) | 1 (1) | 6 (6) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (5) | 2 (4) | 2 (4) | 5 (9) | 0 (0) | 4 (8) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 5 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (3) | 7 (11) | 1 (1) | 1 (1) | 2 (3) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (4) | 1 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (5) | 4 (9) | 6 (6) | 0 (0) | 2 (2) | 2 (2) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 7 (8) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (4) | 2 (3) | 6 (7) | 0 (0) | 2 (3) | 1 (1) | 1 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (4) | 8 (10) | 1 (1) | 3 (4) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 7 (7) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 2 (2) | 3 (3) | 12 (13) | 0 (0) | 4 (9) | 0 (0) | 1 (1)
Peripheral Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (3) | 4 (8) | 4 (4) | 0 (0) | 4 (4) | 1 (1) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea, Exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 7 (7) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (3) | 0 (0) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5) | 4 (6) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 2 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (6) | 6 (9) | 2 (2) | 2 (2) | 6 (6) | 0 (0) | 2 (3) | 1 (1) | 2 (2)
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (5) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rash, Maculo-Papular (Skin and subcutaneous tissue disorders) | 2 (2) | 6 (8) | 4 (5) | 2 (2) | 4 (4) | 0 (0) | 2 (3) | 0 (0) | 2 (2)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 6 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No